CLINICAL TRIAL: NCT04488055
Title: Facilitating Use of the National Suicide Prevention Lifeline in Alcohol Patients
Brief Title: Facilitating Use of the National Suicide Prevention Lifeline in Alcohol Patients (Reach Out)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Mark A. Ilgen, Professor, Department of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00164699; 5R01AA027513-05 (NIH)
Record Dates: First submitted 2020-07-20; First posted 2020-07-27 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Suicide; Alcohol Use Disorder
Keywords: National Suicide Prevention Lifeline
MeSH Terms: conditions — Suicide; Alcoholism

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crisis Line Facilitation (CLF) (Experimental): This single-session intervention addresses the individuals' perceived barriers and facilitators of crisis line use during periods of suicidal crisis.
  Interventions: Behavioral: Crisis Line Facilitation (CLF)
- Enhanced Usual Care (EUC) (Active Comparator): Participants randomized to the EUC condition will receive a brochure (in-person, via email, or via text message) with the NSP Lifeline and a list of outpatient mental health and substance use resources and encouraged to schedule an appointment with a clinical provider if they would like to discuss any current or past symptoms.
  Interventions: Behavioral: Enhanced Usual Care (EUC)

INTERVENTIONS:
Behavioral: Crisis Line Facilitation (CLF) — CLF is a motivational interviewing-based intervention
  Arms: Crisis Line Facilitation (CLF)
Behavioral: Enhanced Usual Care (EUC) — In addition to receiving the brochure, EUC condition participants will meet with a therapist (in-person or remotely) for approximately 15 minutes for a descriptive overview of the brochure.
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
The purpose of this research study is to learn about people who use the National Suicide Prevention (NSP) Lifeline during a suicidal crisis and those who don't. The researchers would also like to learn whether people who have experienced a suicidal crisis could benefit from participating in a therapy session about their thoughts and perceptions of the NSP Lifeline.

ELIGIBILITY:
Inclusion Criteria:

* Probable alcohol use disorder within the past year based on an Alcohol Use Disorders Identification Test (AUDIT) score of 16 or greater
* Report of a suicide attempt within the past year OR a lifetime suicide attempt more than a year ago and current suicide ideation within the past month based on a score of 5 or greater on the Beck Scale for Suicidal Ideation (BSS) or depression in the past month as measured by the Beck Depression Inventory with a of 20 or higher.

Exclusion Criteria:

* Patients who do not understand English
* Prisoners
* Patients with profound psychotic symptoms and/or cognitive deficits that would prevent patients from understanding the content of the intervention and/or assessments.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-17 (Actual)

PRIMARY OUTCOMES:
Crisis line utilization | Up to 12 months
  The Time Line Follow Back (TLFB) assessment will be used as the primary measure of crisis line utilization. Participants will report days of utilization.

SECONDARY OUTCOMES:
Suicidal behavior | Up to 12 months
  The Time Line Follow Back (TLFB) assessment will be the primary measure of suicidal behavior. Participants will report days with suicidal behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ilgen, PhD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Detroit Rescue Mission Ministries, Detroit, Michigan
  - Meridian Health Services, Waterford, Michigan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/55/NCT04488055/ICF_000.pdf